CLINICAL TRIAL: NCT04300738
Title: Evaluation and Comparison of Two Biomarkers (VOP and SCC) for the Prognosis of the Occurrence of Clinical Cardiovascular Events
Acronym: VOP-SCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-A01523-54
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Risk Factor
Keywords: Pulse Wave Velocity; Coronary Calcium Score,; Cardiovascular event,; Cardiovascular risk factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing CT scann for CCS determination (Other)
  Interventions: Device: CCS wit CT Scann measurement

INTERVENTIONS:
Device: CCS wit CT Scann measurement — Measurement with 2 devices
  Other Names: PWV measurement with pOpmètre

SUMMARY:
The aim of our study is to assess the Cardiovascular risk and the quality of the arteries by comparing the Coronary Calcium Score SCC measured with a CT scann and the Pulse Wave Velocity PWV measured with pOpmeter for the prognosis at 6 months of clinical events.

Is there a superiority of PWV compared to SCC:

DETAILED DESCRIPTION:
Two method of cardiovascular risk screening are compared in patient going for Coronary Calcium Score measurement in a outpatient clinic. Ct Scann is expensive, learning time is for at least 2 years, and the reliability is operator dependent.

The Pulse Wave Velocity is measured using a new device with half an hour learning curve, and you get a result within 2 minutes.

1. A non-invasive medical device vs invasive
2. A better benefit-risk ratio
3. A lower diagnostic cost both for equipment and for qualification for use and learning time

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged over 18
2. Any Patient referred to the Bizet Clinic for a CT scan of the coronary arteries
3. Subject affiliated to a social security scheme or beneficiary of such a scheme
4. Lack of participation in another clinical study

Exclusion Criteria:

1. Minor patient
2. Patient with obliterating arterial disease of the lower limbs
3. Patient with Sore fingers and hands
4. Patient with arrhythmia that does not allow measurement of VOP
5. Patient with limb amputation
6. Major subject protected by law, under curatorship or tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Coronary Calcium Score | 12 months
  Coronary Calcium Score,
Pulse Wave Velocity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Benkessou, Paris, France